CLINICAL TRIAL: NCT02408679
Title: A Study to Validate a Predictive Questionnaire for Vitamin D Insufficiency in Healthy Adults
Brief Title: Predictive Questionnaire for Vitamin D Insufficiency in Healthy Adults
Status: Completed | Type: Observational
Sponsor: Lesieur (Industry)
Collaborators: Naturalpha (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-035; ID-RCB Number : 2014-A01633-44 (Other: ANSM)
Record Dates: First submitted 2015-02-05; First posted 2015-04-03 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Healthy Volunteers
Keywords: Vitamin D; Vitamin D Deficiency; Vitamin D Insufficiency; Healthy adults; Predictive questionnaire
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All subjects: 300 eligible subjects will perform a blood sampling for a dosage of serum vitamin D and will fill up a study questionnaire during one visit.
  Interventions: Procedure: Blood sampling; Other: Predictive questionnaire for vitamin D insufficiency

INTERVENTIONS:
Procedure: Blood sampling — One blood sampling will be performed for a serum vitamin D dosage. The volume of blood collected will not exceed 4 ml.
Other: Predictive questionnaire for vitamin D insufficiency — The questionnaire includes 19 questions concerning the following topics : a) sun exposure, b) living situation, c) eating habits and Vitamin D dietary intakes. In addition, two questions will capture demographic data.

SUMMARY:
The purpose of this clinical study is to evaluate the metrological properties of a questionnaire that aims to identify the vitamin D status in reference to a vitamin D blood dosage.

DETAILED DESCRIPTION:
Each subject will perform only one visit (visit V1). The study duration per subject will last about 2 hours. During this visit V1, the subjects will perform a medical exam in order to check their eligibility (general statement and check of inclusion / non-inclusion criteria). The eligible subjects will fill up a study questionnaire and will perform a blood sampling for a dosage of serum vitamin D.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers
* Subject able to communicate with the investigator and the study team, able to read and write and follow all study instructions.
* Written informed consent provided and signed prior screening, after receiving and understanding the subject information.
* Registered with the French Social Security, in agreement with the French law on biomedical experimentation.

Exclusion Criteria:

* Subject with diagnosed osteoporosis, osteopenia or osteomalacia.
* Subject with known disease that contributes in osteoporosis: Rheumatoid arthritis, Malabsorption syndrome, Inflammatory bowel disease, Hyperthyroidism, Hyperparathyroidism.
* Subject with known hepatic impairment.
* Subject with known liver impairment or with a history of renal transplantation.
* Subject with history of cancer.
* Subject with history of bariatric surgery.
* Subject taking or having taken osteoporosis inducing treatment, or treatment with an effect on calcium and phosphorus metabolism during the 3 months prior the visit: Corticosteroids, Enzyme inducing anticonvulsants, Heparin.
* Subject requiring vitamin D supplementation for a diagnosed pathology.
* Pregnant or breastfeeding Female.
* Subject with history of alcohol or drug abuse.
* Participation to any other clinical trial simultaneously and/or not having ended the exclusion period of another clinical trial.
* Subject of legal age unable of giving consent.
* Subject deprived of liberty by judicial or administrative decision.
* Subject of legal age under legal protection.
* Subject having received over 4500 Euros for clinical trial participation within the prior year including the indemnity for the present study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2015-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Questionnaire internal validity | Day 1
  Evaluation of the internal coherence and factorial structure of the questionnaire, establishment of scoring rules
Questionnaire external validity | Day 1
  Prediction of the vitamin D status (threshold value, sensitivity, specificity for vitamin D insufficiency; threshold value, sensitivity, specificity for vitamin D deficiency)
Confounding factors (demographic data) | Day 1
  Interests for coupling the study questionnaire and demographic data (age, gender, Body Mass Index, phototype).

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie BRETON, R&D Innovation Manager, Study Director — Lesieur, France; Xavier Deplanque, MD, Principal Investigator — Clinical Nutrition Center Naturalpha, France
Locations (1):
- Clinical Nutrition Center Naturalpha (CNCN), Lille, France